CLINICAL TRIAL: NCT05758662
Title: The Effect of Subclinical Leaflet Thrombosis and Prosthesis Type on Transcatheter Aortic Valve Degeneration
Brief Title: The Effect of Subclinical Leaflet Thrombosis and Prosthesis Type on Transcatheter Aortic Valve Degeneration (POPular PET TAVI)
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: St. Antonius Research Fund (Unknown); Medtronic (Industry)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, MD, PhD, MSc, St. Antonius Hospital
Other Study IDs: NL82791.100.23
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; TAVR; Subclinical Leaflet Thrombosis; Bioprosthetic Valve Deterioration; Intra-annular; Supra-annular
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-annular: Patients with an intra-annular Sapien TAVI prosthesis
  Interventions: Diagnostic Test: 18F-sodium fluoride Positron Emission Tomography (18F-NaF PET), Cardiac Computed Tomography (CT), Transthoracic Echocardiography (TTE)
- Supra-annular: Patients with a supra-annular CoreValve Evolut TAVI prosthesis
  Interventions: Diagnostic Test: 18F-sodium fluoride Positron Emission Tomography (18F-NaF PET), Cardiac Computed Tomography (CT), Transthoracic Echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: 18F-sodium fluoride Positron Emission Tomography (18F-NaF PET), Cardiac Computed Tomography (CT), Transthoracic Echocardiography (TTE) — Patients undergo a hybrid 18F-NaF-PET CT scan and TTE at five years after TAVI

SUMMARY:
A multicentre cross-sectional cohort study to assess the difference in bioprosthetic micro-calcification activity, detected with 18F-NaF PET-CT, as early marker of transcatheter valve degeneration, between patients with vs. without subclinical leaflet thrombosis at five years after TAVI; and between patients with intra-annular vs. supra-annular TAVI prostheses.

DETAILED DESCRIPTION:
Subclinical leaflet thrombosis (SCLT) occurs frequently after TAVI and has been associated with an increased risk of valve dysfunction. A persistent form of SCLT may lead to thrombus calcification and valve degeneration and increase the long-term risk of symptomatic bioprosthetic valve deterioration. Intra-annular in comparison to supra-annular TAVI valves have been associated with a higher risk of SCLT and valve thrombosis. Intra-annular valves may create larger neo-sinuses and flow stagnation zones, which favour local thrombogenicity. Whether different prosthesis types lead to a higher degree of transcatheter valve calcification and degeneration is currently unexplored. Recently, 18F-sodium fluoride (18F-NaF) positron emission tomography (PET) has emerged as a non-invasive modality capable of imaging bioprosthetic micro-calcification activity, which is an early and powerful predictor of valvular dysfunction and eventually valve failure. In the present study, we investigate for the first time, the differences in quantified bioprosthetic micro-calcification activity with 18F-NaF PET as early marker of transcatheter valve degeneration between patients with and without SCLT and between patients with intra-annular vs. supra-annular prostheses at five years after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Successful TAVI with Sapien or CoreValve Evolut prosthesis about 5 years ago
* Able to undergo hybrid 18F-NaF PET-CT imaging and transthoracic echocardiography
* Written informed consent

Exclusion Criteria:

* Temporary or chronic oral anticoagulation use after TAVI
* Known severe renal insufficiency
* Known severe paravalvular regurgitation
* History of valve-in-valve procedure
* History of aortic valve re-intervention (including percutaneous paravalvular leak closure)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent TAVI about five years ago will be consecutively screened for eligibility from the ongoing, prospective, TAVI registries of the participating study sites and will be asked to undergo hybrid PET-CT imaging and transthoracic echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Quantified bioprosthetic micro-calcification activity | 5 years after TAVI
  18F-NaF uptake originating from any of the bioprosthetic valve leaflets assessed with 18F-NaF Positron Emission Tomography
Subclinical Leaflet Thrombosis | 5 years after TAVI
  Hypo Attenuated Leaflet Thickening (HALT) assessed with cardiac Computed Tomography
Valve dysfunction | 5 years after TAVI
  Transvalvular gradients assessed with transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (4):
- Rigshospitalet, Copenhagen, Denmark
- Netherlands (2):
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Amsterdam UMC, Amsterdam
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Decided upon request